CLINICAL TRIAL: NCT06825793
Title: Clinical Assessment of Semaglutide-Induced Weight Reduction in Obese Populations
Brief Title: Semaglutide's Weight Loss Effects in Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Jia Liu, Director of Endocrinology, Beijing Chao Yang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-Semaglutide-obesity
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLR group (Sham Comparator): Patients with a weight loss of less than 5% at the end of treatment are defined as semaglutide low responders (SLR).
  Interventions: Drug: Semaglutide Subcutaneous Injection
- SHR group (Active Comparator): Patients who experience a weight reduction of ≥15% at the treatment endpoint are defined as high responders to semaglutide (SHR).
  Interventions: Drug: Semaglutide Subcutaneous Injection

INTERVENTIONS:
Drug: Semaglutide Subcutaneous Injection — All subjects received subcutaneous injections of semaglutide over a 28-week treatment period, which included an initial 16-week dose-escalation phase. The escalation protocol began with a starting dose of 0.25 mg administered once weekly. Every 4 weeks, the dose was gradually increased in a stepwise manner to 0.5 mg, 1.0 mg, 1.7 mg, and finally 2.4 mg, each administered once weekly.

SUMMARY:
This is a non-randomized, concurrent, parallel-controlled clinical trial. The objective of this trial is to determine the relationship between weight loss responsiveness to semaglutide in obese patients and their gut microbiota.

DETAILED DESCRIPTION:
Obesity has gradually emerged as a major public health concern. Although the GLP-1 receptor agonist semaglutide is used for chronic weight management in obese patients, significant individual variability exists in its weight-loss efficacy, and the underlying mechanisms remain unclear. Our preliminary studies have revealed that the low-response group to semaglutide exhibits significantly reduced plasma drug concentrations accompanied by a marked increase in the abundance of Prevotella copri (P. copri). Colonization with P. copri was found to attenuate semaglutide's weight-reducing effects in obese mice while decreasing its plasma concentration. In vitro experiments demonstrated an 85% degradation rate of semaglutide after 24-hour co-cultivation with P. copri. Based on these findings, we hypothesize that intestinal P. copri may produce specific enzymes that metabolize semaglutide, thereby influencing its therapeutic efficacy. This project aims to investigate the individual variability in semaglutide response through multi-omics approaches including fecal metagenomic sequencing. Utilizing in vitro bacterial screening platforms combined with gut microbiota gene knockout/heterologous expression systems, protein isolation-activity tracking, and structural characterization, we will elucidate the mechanisms underlying gut microbiota-mediated semaglutide resistance from microbial, animal, and clinical perspectives. The outcomes may identify novel therapeutic targets to overcome semaglutide resistance in weight management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* BMI ≥ 30 kg/m²
* At least one self-reported unsuccessful attempt at lifestyle weight loss

Exclusion Criteria:

* Weight change (self-reported) > 5% in the past 3 months prior to screening
* Use of any medication for obesity indication in the past 3 months prior to screening.
* Use of antidiabetic medications in the past 3 months, or HbA1c ≥ 6.5%, or a history of Type 1 or Type 2 diabetes.
* Use of immunosuppressants, corticosteroids, antidiarrheal drugs, antibiotics, probiotics, lipid-lowering medications, and/or other gastrointestinal motility drugs in the past 3 months prior to screening.
* A history of endocrine-related overweight or obesity diagnoses, such as Cushing's syndrome.
* Triglycerides ≥ 500 mg/dL (5.65 mmol/L) at screening.
* Known clinically significant gastric emptying abnormalities (e.g., severe diabetic gastroparesis or gastric outlet obstruction), gastrointestinal diseases, or surgical history.
* Thyroid dysfunction.
* History of mental illness.
* History or family history of multiple endocrine neoplasia or medullary thyroid cancer, or calcitonin ≥ 6 pg/mL.
* Abnormal liver function at screening, defined as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3*ULN.
* Abnormal kidney function at screening, defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.75m².
* History of cardiovascular disease.
* History of malignancy.
* Pregnancy or breastfeeding.
* Any other physiological, psychological, or other conditions deemed by the investigator as unsuitable for participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | Weight changes will be measured at the following time points: before treatment, and at weeks 4, 8, 12, 16, 20, 24, and 28 after treatment
  When measuring the subject's body weight, ensure shoes, hats, and heavy clothing or accessories are removed, and record the measurement to the nearest 0.1 kg.
Gut microbiota | Gut microtioba will be measured at the following time points: before treatment, and at weeks 4, 8, 12, 16, 20, 24, and 28 after treatment
  Using metagenomic sequencing to assess changes in the composition and abundance of gut microbiota between two groups of subjects. By analyzing the metagenomic data, we will identify specific microbial taxa and functional genes that show significant variation between the groups. This approach will provide insights into the microbial diversity, stability, and metabolic capabilities of the gut microbiome.

SECONDARY OUTCOMES:
Blood biochemical indicators | Blood biochemical indicators will be measured at the following time points: before treatment, and at weeks 16 and 28 after treatment
  The study subjects were all in a fasting state. A professional nurse collected 1 tube of blood from the antecubital vein, and the blood sample was sent to the hospital's laboratory for testing on the same morning. The tests included complete blood count, fasting blood glucose, fasting insulin, glycated hemoglobin, serum triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, alanine aminotransferase (ALT), uric acid, creatinine, electrolytes, and other measurements. All tests were conducted using an automatic biochemical analyzer. Post-test blood was used to measure serum DPP4 concentration and GLP-1 activity, among others.
The blood concentration of semaglutide | concentration of semaglutide will be measured at weeks 24 after treatment
  At 24 weeks, all study subjects had one tube of blood collected from the antecubital vein in a fasting state by a professional nurse. After centrifugation, the plasma was collected and analyzed for semaglutide plasma drug concentration using liquid chromatography-tandem mass spectrometry (LC-MS/MS).
BMI | BMI will be measured at the following time points: before treatment, and at weeks 4, 8, 12, 16, 20, 24, and 28 after treatment
  Height (measured without shoes, accurate to 0.1 cm), weight (measured without shoes, hat, heavy clothing, and accessories, accurate to 0.1 kg), and Body Mass Index (BMI) are calculated after converting the height unit. BMI = weight / height² (kg/m²).

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, Study Chair — Beijing Chao Yang Hospital